CLINICAL TRIAL: NCT07153731
Title: Observation on the Clinical Efficacy of Shenkangling in the Treatment of Renal Ischemia-reperfusion Injury (Kidney Deficiency and Blood Stasis Syndrome)
Brief Title: The Clinical Research of Traditional Chinese Medicine Compound Formulas
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-042
Record Dates: First submitted 2025-05-11; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Urologic Injuries; Urology
Keywords: Traditional Chinese Medicine; Renal Fibrosis; Renal Ischemia-reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): No treatment
- Shenkangling group (Experimental): Shenkangling
  Interventions: Drug: Shenkangling

INTERVENTIONS:
Drug: Shenkangling — Chinese herbal tonics taken orally: Shenkangling, one dose, 2 times a day, 1 time before breakfast and 1 time 30 minutes after dinner.
  Arms: Shenkangling group

SUMMARY:
To observe the efficacy and safety of Shenkangling, a traditional Chinese medicine decoction, for renal ischemia-reperfusion injury, and to provide evidence-based medical evidence and ideas for clinical therapeutic use.

DETAILED DESCRIPTION:
1. Study Design and Methods 1.1 Research Method A multicenter, open-label study design is employed. 1.2 Source of Participants Clinical observation cases are from patients with ischemia-reperfusion injury caused by partial nephrectomy or renal exploration, admitted between March 2025 and December 2026 to the Department of Urology at Zhejiang University School of Medicine Fourth Affiliated Hospital and Fujian University of Traditional Chinese Medicine Affiliated People's Hospital. A total of 100 subjects are included.

1.3 Participant Selection and Exclusion Criteria 1.3.1 Western Medicine Diagnostic Criteria

1. Partial nephrectomy due to renal tumor: Based on the "Chinese Expert Consensus on Laparoscopic and Robotic Partial Nephrectomy for Renal Tumors," the general diagnosis of renal tumor should be met, with the maximum tumor diameter ≤ 4 cm, and the indication for partial nephrectomy.
2. Partial nephrectomy due to renal cyst: Based on the "Consensus on the Safety of Surgical Treatment for Simple Renal Cysts," the general diagnosis of renal cyst should be met, and partial nephrectomy should be indicated.
3. Partial nephrectomy or renal exploration due to renal injury: According to the "Urological Injury Diagnosis and Treatment Guidelines" issued by the Chinese Urological Association, injuries such as renal contusion, partial renal laceration, complete renal laceration, and renal pedicle injury caused by open or closed trauma, which are indications for partial nephrectomy or renal exploration.
4. Partial nephrectomy due to renal hamartomas, complex renal cysts, or other conditions: Based on the "2022 Edition of the China Urological and Andrological Diseases Diagnosis and Treatment Guidelines," the general diagnosis of these diseases should be met, and partial nephrectomy should be indicated.

1.3.2 Traditional Chinese Medicine Diagnostic Criteria

Based on clinical manifestations and the "Guidelines for Clinical Research on New Chinese Medicines" and "General Principles for Clinical Research on New Chinese Medicines" established by the People's Republic of China, and referring to the opinions of various scholars, the criteria are as follows:

Kidney Deficiency and Blood Stasis Syndrome Main Symptoms: Low back and spine soreness or stabbing pain or fixed pain, fatigue, swelling, susceptibility to colds, afternoon fever, palms and soles of the feet hot, dark or dull complexion.

Secondary Symptoms: Dry mouth, dry throat, dark red throat, skin and nails rough or numb limbs, tongue red or slightly red, or tongue purple and dark with bruises or spots, thin pulse.

At least one main symptom and at least two secondary symptoms must be present, with tongue and pulse findings consistent.

1.3.3 Inclusion Criteria

1. Meets the Western medical diagnostic criteria, requiring renal ischemia-reperfusion surgery with renal artery occlusion time ≤ 30 minutes;
2. Meets the Traditional Chinese Medicine syndrome differentiation criteria;
3. Age between 18 and 65 years;
4. Voluntary participation and signing of informed consent. 1.3.4 Exclusion Criteria

(1) Patients with stage 4 or 5 renal failure or acute renal failure; (2) Diagnosed with systemic lupus erythematosus, drug-induced kidney damage, or other secondary causes; (3) Not meeting the diagnosis of renal ischemia-reperfusion injury; (4) Not within the scope of the drug's effect; (5) Long-term use of other related drugs, such as those on long-term oral Chinese medicines like Jin Kui Shen Qi Wan, or unable to stop the medication immediately; (6) Severe deformities, disabilities, or loss of work ability; (7) Co-existing severe primary diseases such as heart, brain, liver, hematological, or endocrine system diseases, and psychiatric disorders; (8) Pregnant or breastfeeding women; (9) Critically ill patients; (10) Other conditions deemed unsuitable for inclusion by the researchers. 1.3.5 Participant Withdrawal 1.3.5.1 Investigator-Determined Withdrawal

1. The investigator determines that it is necessary to stop the study from an ethical perspective;
2. Serious adverse events occur, and the participant should no longer continue the trial;
3. Serious co-morbidities arise during treatment;
4. The investigator determines that withdrawal from the study is in the participant's best interest;
5. Other reasons. 1.3.5.2 Participant-Determined Withdrawal Participants have the right to withdraw from the trial at any stage, or if the participant does not withdraw informed consent but fails to continue medication or follow-up, they are considered lost to follow-up.

1.3.6 Dropout Criteria

1. Serious adverse events or complications occur;
2. The participant requests to withdraw from the trial during the study;
3. Unable to contact the participant during the trial. 1.3.7 Exclusion Criteria

(1) Found to not meet inclusion criteria after enrollment; (2) Poor compliance with the study protocol, including not following prescribed medication or clinical tests; (3) Incomplete data during the trial, making it impossible to evaluate the drug's efficacy and safety.

2.4 Treatment Plan and Grouping 2.4.1 Trial Medication Shenkangling Composition: Astragalus, Rehmannia, Cornus, Dioscorea, Poria, Moutan Root Bark, Panax Notoginseng, etc.

Formulation: Decoction Dosage: 150 ml per dose Source: Zhejiang Sanxi Tang Chinese Medicine Co., Ltd. 2.4.2 Grouping This study involves two groups: Patients are randomly divided into the control group and experimental group, each with 40 cases. The control group receives standard treatment (post-operative anti-infection, fluid supplementation, and symptomatic treatment), while the experimental group receives Shenkangling decoction orally on top of standard treatment (one dose per day, split into two doses: one 30 minutes before breakfast and one 30 minutes after dinner).

Randomization Method: Random numbers (1-96) are generated using SPSS software and randomly assigned to the Shen Kang Ling group and the control group, each receiving 48 numbers. The distribution results are kept confidential by the group leader, who determines and records the grouping and sequence number of patients.

2.5 Statistical Analysis Method SPSS v22.0 will be used for statistical analysis. Categorical data will be analyzed using the χ² test. Continuous data will be presented as means ± standard deviations (SD) and compared using t-tests. Statistical significance is set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfillment of western medical diagnostic criteria requiring renal ischemia-reperfusion surgical operation and renal artery clamping time ≤ 30 min
2. Meets the criteria for Chinese medicine identification
3. 18 ≤ age ≤ 65
4. Voluntary participation with signed informed consent

Exclusion Criteria:

1. Patients with stage 4 or 5 renal insufficiency or patients with acute renal failure
2. Those with secondary factors such as systemic lupus erythematosus, drug-induced renal damage, etc. confirmed by examination
3. Does not meet the diagnosis of renal ischemia-reperfusion injury
4. Cases not within the scope of action of the drug
5. Those who have been taking other related therapeutic drugs for a long period of time, e.g., taking Chinese medicines such as Jingui Shenqi Pills by mouth for a long period of time, or those who are unable to stop taking the medicines immediately.
6. Advanced deformity, disability, loss of labor force
7. Combined heart, brain, liver, hematopoietic system, endocrine system and other serious primary diseases and psychiatric patients
8. Pregnant or lactating women
9. Critically ill patients
10. Other circumstances deemed inappropriate for inclusion in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of 24-hour urine protein excretion | From enrollment to the end of treatment at 8 weeks
Levels of renal function | From enrollment to the end of treatment at 8 weeks
  Biochemical tests for blood creatinine and urea nitrogen
Specific gravity of urine | From enrollment to the end of treatment at 8 weeks
blood viscosity | From enrollment to the end of treatment at 8 weeks
  By measuring the flow rate of blood in capillaries to evaluate blood viscosity
Levels of renal fibrosis（CⅣ、PCⅢ、CTGF、TIMP-1） | From enrollment to the end of treatment at 8 weeks
Levels of electrolytes | From enrollment to the end of treatment at 8 weeks
  Mainly includes the following indicators: Potassium ion, Sodium ion, Chloride ion, Calcium ions.
Levels of urobilinogen | From enrollment to the end of treatment at 8 weeks
Occult blood in urine | From enrollment to the end of treatment at 8 weeks
White blood cell count of urine | From enrollment to the end of treatment at 8 weeks
Red blood cell count of urine | From enrollment to the end of treatment at 8 weeks
Levels of urine NAG enzyme | From enrollment to the end of treatment at 8 weeks
Levels of urine β2-microglobulin | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No